CLINICAL TRIAL: NCT00019409
Title: A Randomized Study of Two Methods of CNS Prophylaxis in Patients With Acute Lymphoblastic Leukemia
Brief Title: Radiation Therapy to the Head or Intrathecal Chemotherapy Plus High Dose Cytarabine in Preventing CNS Disease in Children With Acute Lymphoblastic Leukemia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 999998007; 98-C-N007; MCP943; NCI-0H98-C-N007; CDR0000066120
Record Dates: First submitted 2001-07-11; First posted 2004-02-27 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Leukemia
Keywords: untreated childhood acute lymphoblastic leukemia; childhood acute lymphoblastic leukemia in remission; L1 childhood acute lymphoblastic leukemia; L2 childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Mercaptopurine; Methotrexate; Prednisone; Hydrocortisone; Vincristine; Radiotherapy

INTERVENTIONS:
Drug: asparaginase
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: mercaptopurine
Drug: methotrexate
Drug: prednisone
Drug: therapeutic hydrocortisone
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Giving radiation therapy to the head or intrathecal chemotherapy may prevent cancer cells from spreading to the brain. It is not yet known which treatment regimen is more effective for acute lymphoblastic leukemia.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy to the head or intrathecal chemotherapy plus high dose cytarabine in preventing CNS disease in children who have acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy and toxicity of cranial radiation vs triple intrathecal chemotherapy plus high dose systemic cytarabine for prophylaxis of CNS disease in children with acute lymphoblastic leukemia. II. Compare the overall survival rates of these patients after these treatments.

OUTLINE: This is a randomized, multicenter study for approved centers in India only. All patients receive induction therapy and then are randomized to one of two treatment arms. Patients assigned to arm I receive high dose cytarabine and no cranial radiation and patients assigned to arm II receive cranial radiation and no high dose cytarabine. Induction 1: Patients receive vincristine IV on days 1, 8, 15, 22, and 29, oral prednisone on days 1-28, triple intrathecal therapy (methotrexate, hydrocortisone, and cytarabine; TIT) on days 1, 8, 15, and 22, asparaginase IM every other day on days 2-20, and daunorubicin IV on days 8, 15, and 29. Patients who achieve remission proceed to randomization. Arm I: Induction 2: Patients receive oral mercaptopurine daily on days 1-7 and 22-28, cytarabine IV over 3 hours every 12 hours for 4 doses on days 1-2 and 22-23, cyclophosphamide IV on days 1 and 22, and TIT on days 8 and 29. Induction 1 is repeated, then patients proceed to consolidation when blood counts have recovered sufficiently. Consolidation: Induction 2 is repeated, then patients proceed to maintenance when blood counts have recovered sufficiently. Maintenance 1: Patients receive vincristine IV and daunorubicin IV on day 1; oral prednisone on days 1-7; asparaginase IM on days 1, 3, 5, and 7; oral methotrexate once a week beginning on day 15 and skipping every 4th week, for a total of 12 weeks; oral mercaptopurine beginning on day 15 for 3 weeks out of 4, for a total of 12 weeks; and TIT on days 1 and 36. Maintenance 2: Patients receive cytarabine IV over 3 hours every 12 hours for 4 doses on days 1-2, cyclophosphamide IV over 30 minutes on day 1, and methotrexate, mercaptopurine, and TIT on days 8 and 36. A total of 6 maintenance courses are administered, alternating maintenance 1 and 2. Arm II: Induction 2: Patients receive oral mercaptopurine daily on days 1-7 and 15-21, cyclophosphamide IV over 30 minutes on days 1 and 15, and intrathecal methotrexate on days 1, 8, 15, and 22. Patients then receive cranial radiation daily on days 4-12. Induction 1 is repeated, then patients proceed to consolidation after blood counts have recovered sufficiently. Consolidation: Patients receive cyclophosphamide IV over 30 minutes on days 1-15, vincristine IV on days 1 and 15, oral mercaptopurine daily on days 1-7 and 15-21, and cytarabine subcutaneously every 12 hours for 6 doses on days 1-3 and 15-17. Patients proceed to maintenance when blood counts recover sufficiently. Maintenance: Same as maintenance 1 in arm I, excluding TIT. A total of 6 courses are administered. All patients are followed monthly for the first 6 months, then every other month for the next 6 months, every 3 months for the next 2 years, every 6 months for the next 5 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 1100 patients (550 per arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Cytologically confirmed acute lymphoblastic leukemia Greater than 25% lymphoblasts in bone marrow No mediastinal or localized lymphoblastic lymphoma No single node or extranodal site without bone marrow involvement No B cell lymphoma (Burkitt's or L3 FAB) No blast cells positive for myeloperoxidase No CNS disease

PATIENT CHARACTERISTICS: Age: 1-20 Performance status: Not specified Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: Not specified Renal: Not specified Other: HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: No prior corticosteroids Radiotherapy: No prior radiotherapy Surgery: Not specified

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 1999-10; Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Trevor Magrath, MD, FRCP, FRCPath, Study Chair — National Cancer Institute (NCI)
Locations (6):
- United States (2):
  - Pediatric Oncology Branch, Bethesda, Maryland
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
- India (4):
  - Kidwai Memorial Institute of Oncology, Bangalore
  - Cancer Institute (W.I.A.), Madras
  - Tata Memorial Centre, Mumbai
  - All-India Institute of Medical Sciences, New Delhi